CLINICAL TRIAL: NCT05307679
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety, Efficacy, and Pharmacodynamics of 52 Weeks of Treatment With Basmisanil in Participants Aged 2 to 14 Years Old With Dup15q Syndrome Followed by a 2-Year Optional Open-Label Extension
Brief Title: A Study to Evaluate the Safety and Efficacy of Basmisanil Treatment in Children Aged 2-14 Years With Dup15q Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to sponsor decision and not related to safety or tolerability.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP42992
Record Dates: First submitted 2022-03-25; First posted 2022-04-01 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Dup15q Syndrome
Keywords: dup15q; dup15q syndrome; 15q; duplication 15q; 15q duplication; chromosome 15q duplication; 15q duplication syndrome; duplication 15; triplication 15
MeSH Terms: conditions — Polyposis Syndrome, Hereditary Mixed, 1; Chromosome 15q, trisomy | interventions — basmisanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Basmisanil (Experimental): Participants will receive oral basmisanil twice daily (BID) on the first day of treatment, then three times per day (TID) until the end of Part 1 of the trial (Day 365) or the end of Part 2 (Day 1095)
  Interventions: Drug: Basmisanil
- Placebo (Placebo Comparator): Participants will receive oral placebo BID on the first day of treatment, then TID until the end of Part 1 of the trial (Day 365).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Basmisanil — Participants will receive oral basmisanil at age-appropriate dosages
  Arms: Basmisanil
Drug: Placebo — Participants will receive oral placebo
  Arms: Placebo

SUMMARY:
This study consists of two parts. Part 1 will evaluate the safety, efficacy, and pharmacodynamics of 52-weeks of basmisanil treatment in children and adolescents (aged 2-14 years) with Dup15q syndrome. Part 1 will test the hypothesis that negative allosteric modulation of a GABAA receptor subtype can address excessive receptor function and positively impact core neurodevelopmental disease feature in individuals with Dup15q syndrome. Part 2 is an optional 2-year open-label extension to evaluate long-term safety, tolerability, and to provide supportive evidence of benefit of continued treatment with basmisanil in selected efficacy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Documented maternal duplication (3 copies) or triplication (4 copies) of the chromosome 15q11.2-q13.1 region that includes the Prader Willi/Angelman critical region defined as [BP2-BP3] segment
* Dup15q syndrome Clinician Global Impression of Severity scale (Dup15q CGI-S) overall severity score ≥ 4 (at least moderately ill)
* Body weight equal to or above the third percentile for age
* Participant has a parent, caregiver, or legally authorized representative (hereinafter "caregiver") of at least 18 years of age, who is fluent in the local language at the site, and capable and willing to provide written informed consent for the participant, according to International Council for Harmonisation and local regulations
* Participant's caregiver must be living with the participant and, in the opinion of the Investigator, able and willing to reliably assess the participant's ongoing condition, to accompany the participant to all clinic visits, and ensure compliance to study treatment throughout the study. The same caregiver is able and willing to complete the caregiver assessments and is available to the Investigational Site by telephone or email if needed
* Participant's caregiver is able and willing to use electronic devices to record information on the participant's condition and to complete assessments at home and agrees to home nursing visits, if local regulations allow for it and if home nursing service is available in the country/region

Exclusion Criteria:

* Uncontrolled epilepsy at screening (as defined by the protocol)
* Lymphoma, leukemia, or any malignancy within the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Clinically significant ECG abnormalities at Screening
* Clinically significant abnormalities in laboratory test results at screening (including positive results for HIV, hepatitis B and/or hepatitis C)
* Allowed prior existing medication should be on a stable regimen (or frequency of intervention) for at least 6 weeks, and at least 8 weeks for anti-epileptic treatment, prior to Screening
* Non-pharmacological / behavioral therapies should not be stopped or newly started at least 6 weeks prior to Screening and are expected to remain stable for the entire study duration (excluding changes related to standard age and educational interventional programs and minor interruptions such as illness or vacation
* Concomitant use of prohibited medications
* Participation in an investigational drug study within one month or within 6 × the elimination half-life, whichever is longer, prior to dosing in the study
* Significant risk for suicidal behavior, as assessed through the suicidal behavior question adapted from the Columbia Classification Algorithm for Suicide Assessment (C-CASA) (participants ≥ 6 years of age only)
* Known sensitivity to any of the study treatments or components thereof or drug or other allergy that, in the opinion of the Investigator, contraindicates the participation in the study, including severe lactose intolerance (e.g., unable to tolerate 250 mL [8 oz. or 1 cup] of milk, ice cream, or yogurt)
* Concomitant clinically relevant disease or condition or any clinically significant finding at screening that could interfere with, or for which, the treatment might interfere with, the conduct of the study or that would pose an unacceptable risk to the participants in this study
* Known active or uncontrolled bacterial, viral, or other infection (excluding fungal infections of nail beds) or any major clinically significant episode of infection or hospitalization (relating to the completion of the course of antibiotics) within 6 weeks prior to the start of drug administration

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
- Spain (2):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital Universitario La Paz, Madrid
- Evelina London Children's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- See also: https://forpatients.roche.com/ — https://forpatients.roche.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Part 1: Participants received oral placebo twice (BID) on the first day of treatment, then three times daily (TID) to Day 365.
- Basmisanil: Part 1: Participants received oral basmisanil BID on the first day of treatment, then TID to Day 365.
  Part 2: Participants who completed Part 1 were to receive oral basmisanil for approximately 2 years.
Period: Overall Study
Arm/Group | Placebo | Basmisanil
Started | 2 | 5
Completed | 0 | 0
Not Completed | 2 | 5
Not completed — Study terminated by sponsor or physician decision | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Basmisanil | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.0 (1.4) | 8.8 (2.2) | 8.6 (1.9)
Sex/Gender, Customized [Number; unit: Count of Participants]
  Female + Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants were not consented on the collection of race and ethnicity data.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants were not consented on the collection of race and ethnicity data.

OUTCOME MEASURES:

1. Primary Outcome: Vineland-3 Adaptive Behavior Scales, 3rd Edition Composite Scores
Description: The Vineland-3 is an instrument that measures communication, daily living skills, socialization, and motor skills for those with intellectual and developmental disabilities. Items consist of open-ended questions related to activities and behavior and are scored as 2 = Usually, 1 = Sometimes, and 0 = Never. Items requiring a binary response are scored as 2 = Yes, 0. Standard scores for the adaptive behavior composite range from 20-160; lower scores indicate lower adaptive functioning.
Time Frame: Baseline, Day 183, Day 365
Population: ITT population: All randomized participants who received ≥1 dose. Participants were allocated to the treatment arm they were randomized to.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Baseline | 30.50 [30.0 to 31.0] | 36.00 [27.0 to 52.0]
  Day 183: number analyzed (Participants) | 1 | 1
  Day 183 | 28.00 [28.0 to 28.0] | 32.00 [32.00 to 32.00]
  Day 365: number analyzed (Participants) | 1 | 0
  Day 365 | 32.00 [32.00 to 32.00] |

2. Secondary Outcome: Vineland-3 Gross and Fine Motor Subdomains Scores
Description: The Vineland-3 is an instrument that measures communication, daily living skills, socialization, and motor skills for those with intellectual and developmental disabilities. Items consist of open-ended questions related to activities and behavior and are scored as 2 = Usually, 1 = Sometimes, and 0 = Never. Items requiring a binary response are scored as 2 = Yes, 0. V-scale scores for the gross and fine motor domains range from 1-24; lower scores indicate lower adaptive functioning.
Time Frame: Baseline, Day 183, Day 365
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 2
Units on a scale
  Gross Motor V-Scale Score - Baseline | 1.00 [1.0 to 1.0] | 4.50 [1.0 to 8.0]
  Gross Motor V-Scale Score - Day 183: number analyzed (Participants) | 1 | 0
  Gross Motor V-Scale Score - Day 183 | 4.00 [4.00 to 4.00] |
  Gross Motor V-Scale Score - Day 365: number analyzed (Participants) | 1 | 0
  Gross Motor V-Scale Score - Day 365 | 1.00 [1.0 to 1.0] |
  Fine Motor V-Scale Score - Baseline | 1.00 [1.0 to 1.0] | 3.00 [1.0 to 5.0]
  Fine Motor V-Scale Score - Day 183: number analyzed (Participants) | 1 | 0
  Fine Motor V-Scale Score - Day 183 | 1.00 [1.00 to 1.00] |
  Fine Motor V-Scale Score - Day 365: number analyzed (Participants) | 1 | 0
  Fine Motor V-Scale Score - Day 365 | 1.00 [1.00 to 1.00] |

3. Secondary Outcome: Vineland 3 Expressive and Receptive Communication Subdomains
Description: The Vineland-3 is an instrument that measures communication, daily living skills, socialization, and motor skills for those with intellectual and developmental disabilities. Items consist of open-ended questions related to activities and behavior and are scored as 2 = Usually, 1 = Sometimes, and 0 = Never. Items requiring a binary response are scored as 2 = Yes, 0. V-scale scores for the expressive and receptive communication subdomains range from 1-24; lower scores indicate lower adaptive functioning.
Time Frame: Baseline, Day 183, Day 365
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Expressive Communication V-Scale Score - Baseline | 1.00 [1.0 to 1.0] | 1.00 [1.0 to 11.0]
  Expressive Communication V-Scale Score - Day 183: number analyzed (Participants) | 1 | 1
  Expressive Communication V-Scale Score - Day 183 | 1.00 [1.0 to 1.0] | 1.00 [1.0 to 1.0]
  Expressive Communication V-Scale Score - Day 365: number analyzed (Participants) | 1 | 0
  Expressive Communication V-Scale Score - Day 365 | 1.00 [1.0 to 1.0] |
  Receptive Communication V-Scale Score - Baseline | 1.00 [1.0 to 1.0] | 1.00 [1.0 to 6.0]
  Receptive Communication V-Scale Score - Day 183: number analyzed (Participants) | 1 | 1
  Receptive Communication V-Scale Score - Day 183 | 1.00 [1.0 to 1.0] | 1.00 [1.0 to 1.0]
  Receptive Communication V-Scale Score - Day 365: number analyzed (Participants) | 1 | 0
  Receptive Communication V-Scale Score - Day 365 | 1.00 [1.0 to 1.0] |

4. Secondary Outcome: Vineland-3 Play and Leisure Time and Interpersonal Relationships Subdomains
Description: The Vineland-3 is an instrument that measures communication, daily living skills, socialization, and motor skills for those with intellectual and developmental disabilities. Items consist of open-ended questions related to activities and behavior and are scored as 2 = Usually, 1 = Sometimes, and 0 = Never. Items requiring a binary response are scored as 2 = Yes, 0. V-scale scores for the play and leisure time, and interpersonal relationships subdomains range from 1-24; lower scores indicate lower adaptive functioning.
Time Frame: Baseline, Day 153, Day 365
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Play and Leisure V-Scale Score - Baseline | 1.00 [1.0 to 1.0] | 1.00 [1.0 to 9.0]
  Play and Leisure V-Scale Score - Day 183: number analyzed (Participants) | 1 | 1
  Play and Leisure V-Scale Score - Day 183 | 1.00 [1.0 to 1.0] | 1.00 [1.0 to 1.0]
  Play and Leisure V-Scale Score - Day 365: number analyzed (Participants) | 1 | 0
  Play and Leisure V-Scale Score - Day 365 | 1.00 [1.0 to 1.0] |
  Interpersonal Relationships V-Scale Score - Baseline | 1.50 [1.0 to 2.0] | 1.00 [1.0 to 9.0]
  Interpersonal Relationships V-Scale Score - Day 183: number analyzed (Participants) | 1 | 1
  Interpersonal Relationships V-Scale Score - Day 183 | 3.00 [3.0 to 3.0] | 1.00 [1.0 to 1.0]
  Interpersonal Relationships V-Scale Score - Day 365: number analyzed (Participants) | 1 | 0
  Interpersonal Relationships V-Scale Score - Day 365 | 3.00 [3.0 to 3.0] |

5. Secondary Outcome: Mullen Scales of Early Learning (MSEL) Gross and Fine Motor Domains
Description: The MSEL are designed for a certified rater to provide an assessment of cognitive ability and motor development of typically developing children from birth through age 68 months. It was administered to all participants in this study irrespective of their chronological age. The instrument consists of 124 items across five scales measuring Gross Motor, Visual Reception, Fine Motor, Expressive Language, and Receptive Language. Each item is scored from 0-5 points with total raw score ranges of 0-100 (gross motor) and 0-78 (fine motor). Lower score indicate lower developmental abilities; higher scores indicate greater developmental abilities.
Time Frame: Baseline, Day 183, Day 365
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Gross Motor - Baseline | 20.50 [14.0 to 27.0] | 19.00 [13.0 to 35.0]
  Gross Motor - Day 183: number analyzed (Participants) | 1 | 1
  Gross Motor - Day 183 | 24.00 [24.0 to 24.0] | 18.00 [18.0 to 18.0]
  Gross Motor - Day 365: number analyzed (Participants) | 1 | 0
  Gross Motor - Day 365 | 1.00 [1.0 to 1.0] |
  Fine Motor - Baseline | 15.50 [13.0 to 18.0] | 15.00 [6.0 to 30.0]
  Fine Motor - Day 183: number analyzed (Participants) | 1 | 1
  Fine Motor - Day 183 | 18.00 [18.0 to 18.0] | 9.00 [9.0 to 9.0]
  Fine Motor - Day 365: number analyzed (Participants) | 1 | 0
  Fine Motor - Day 365 | 11.00 [11.0 to 11.0] |

6. Secondary Outcome: MSEL Visual Reception Domain Scores
Description: The MSEL are designed for a certified rater to provide an assessment of cognitive ability and motor development of typically developing children from birth through age 68 months. It was administered to all participants in this study irrespective of their chronological age. The instrument consists of 124 items across five scales measuring Gross Motor, Visual Reception, Fine Motor, Expressive Language, and Receptive Language. Each item is scored from 0-5 points with a total raw score range of 0-50. Lower score indicate lower developmental abilities; higher scores indicate greater developmental abilities.
Time Frame: Baseline, Day 183
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Baseline | 14.00 [11.0 to 17.0] | 4.00 [2.0 to 42.0]
  Day 183: number analyzed (Participants) | 1 | 1
  Day 183 | 21.00 [21.0 to 21.0] | 5.00 [5.0 to 5.0]
  Day 365: number analyzed (Participants) | 1 | 0
  Day 365 | 13.00 [13.0 to 13.0] |

7. Secondary Outcome: MSEL Expressive and Receptive Language Subdomains
Description: The MSEL are designed for a certified rater to provide an assessment of cognitive ability and motor development of typically developing children from birth through age 68 months. It was administered to all participants in this study irrespective of their chronological age. The instrument consists of 124 items across five scales measuring Gross Motor, Visual Reception, Fine Motor, Expressive Language, and Receptive Language. Each item is scored from 0-5 points with a total raw score range of 0-50 (expressive language) or 0-48 (receptive language). Lower score indicate lower developmental abilities; higher scores indicate greater developmental abilities.
Time Frame: Baseline, Day 183
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Expressive Language - Baseline | 12.50 [12.0 to 13.0] | 17.00 [6.0 to 29.0]
  Expressive Language - Day 183: number analyzed (Participants) | 1 | 1
  Expressive Language - Day 183 | 23.00 [23.0 to 23.0] | 6.00 [6.0 to 6.0]
  Expressive Language - Day 365: number analyzed (Participants) | 1 | 0
  Expressive Language - Day 365 | 7.00 [7.0 to 7.0] |
  Receptive Language - Baseline | 10.00 [7.0 to 13.0] | 16.00 [9.0 to 28.0]
  Receptive Language - Day 183: number analyzed (Participants) | 1 | 1
  Receptive Language - Day 183 | 17.00 [17.0 to 17.0] | 11.00 [11.0 to 11.0]
  Receptive Language - Day 365: number analyzed (Participants) | 1 | 0
  Receptive Language - Day 365 | 13.00 [13.0 to 13.0] |

8. Secondary Outcome: Dup15q Syndrome Clinician Global Impression of Severity (CGI-S) Scale Scores
Description: The Dup15q CGI-S is a 10-domain clinician-rated measure on a 6-point scale that measures global severity of illness at a given point in time. The ten domains are seizures, expressive communication difficulties, fine motor skills difficulties, gross motor skills difficulties, cognitive/intellectual impairment, impairment in activities of daily living/self-care, socialization, maladaptive behavior, sleep difficulties, and overall severity. Response options are 1-none, 2-very mild, 3-mild, 4-moderate, 5-severe, and 6-very severe.
Time Frame: Baseline until Day 395, or early termination (prior to Day 395)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Baseline | 4.00 [4.0 to 4.0] | 4.00 [4.0 to 6.0]
  Day 28 | 4.00 [4.0 to 4.0] | 4.00 [3.0 to 6.0]
  Day 92: number analyzed (Participants) | 1 | 3
  Day 92 | 4.00 [4.0 to 4.0] | 4.00 [4.0 to 6.0]
  Day 183: number analyzed (Participants) | 1 | 1
  Day 183 | 4.00 [4.0 to 4.0] | 4.00 [4.0 to 4.0]
  Day 274: number analyzed (Participants) | 1 | 0
  Day 274 | 4.00 [4.0 to 4.0] |
  Day 365: number analyzed (Participants) | 1 | 0
  Day 365 | 4.00 [4.0 to 4.0] |
  Follow-Up Day 395: number analyzed (Participants) | 0 | 3
  Follow-Up Day 395 |  | 5.00 [4.0 to 6.0]
  Early Termination: number analyzed (Participants) | 0 | 1
  Early Termination |  | 6.00 [6.0 to 6.0]

9. Secondary Outcome: Dup15q Syndrome Clinician Global Impression of Change Scale (CGI-C) Scores
Description: The Dup15q CGI-C is a 10-domain clinician-rated measure on a 7-point scale that assesses the clinician's impression of change in illness compared with baseline. The ten domains are seizures, expressive communication difficulties, fine motor skills difficulties, gross motor skills difficulties, cognitive/intellectual impairment, impairment in activities of daily living/self-care, socialization, maladaptive behavior, sleep difficulties, and overall severity. Response options are 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse. The CGI does not yield a global score.
Time Frame: Day 28 - Day 395 or early termination (prior to Day 395)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Day 28: number analyzed (Participants) | 2 | 4
  Day 28 | 3.50 [3.0 to 4.0] | 3.00 [2.0 to 3.0]
  Day 92: number analyzed (Participants) | 1 | 3
  Day 92 | 3.00 [3.0 to 3.0] | 3.00 [2.0 to 4.0]
  Day 183: number analyzed (Participants) | 1 | 1
  Day 183 | 4.00 [4.0 to 4.0] | 3.00 [3.0 to 3.0]
  Day 274: number analyzed (Participants) | 1 | 0
  Day 274 | 4.00 [4.0 to 4.0] |
  Day 365: number analyzed (Participants) | 1 | 0
  Day 365 | 3.00 [3.0 to 3.0] |
  Follow-Up Day 395: number analyzed (Participants) | 0 | 3
  Follow-Up Day 395 |  | 3.00 [3.0 to 4.0]
  Early Termination: number analyzed (Participants) | 0 | 1
  Early Termination |  | 4.00 [4.0 to 4.0]

10. Secondary Outcome: Aberrant Behavior Checklist - Second Edition - Community Version (ABC-2-C) Domain Scores - Irritability
Description: The ABC-2 is an updated, empirically derived, validated 58-item caregiver-completed rating scale that measures the severity of a range of maladaptive behaviors commonly observed in children, adolescents, and adults with intellectual and developmental disabilities. The Community version of the scale (ABC-2-C) will be used. It is designed for use in individuals who are not residing in institutional settings. The checklist assesses symptoms across five domains: irritability, social withdrawal, stereotypic behavior, hyperactive/noncompliance, and inappropriate speech. Items are scored on a 4-point scale from 0 (never) to 3 (severe problem). The irritability domain score range is 0-45, with higher score indicating greater severity.
Time Frame: Baseline - Day 365, or early termination (prior to Day 365)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Baseline | 11.00 [11.0 to 11.0] | 15.00 [3.0 to 40.0]
  Day 28: number analyzed (Participants) | 2 | 3
  Day 28 | 10.00 [6.0 to 14.0] | 15.00 [5.0 to 18.0]
  Day 92: number analyzed (Participants) | 1 | 3
  Day 92 | 17.00 [17.0 to 17.0] | 16.00 [5.0 to 23.0]
  Day 183: number analyzed (Participants) | 1 | 1
  Day 183 | 20.00 [20.0 to 20.0] | 28.00 [28.0 to 28.0]
  Day 274: number analyzed (Participants) | 1 | 0
  Day 274 | 16.00 [16.0 to 16.0] |
  Day 365: number analyzed (Participants) | 1 | 0
  Day 365 | 13.00 [13.0 to 13.0] |
  Early Termination: number analyzed (Participants) | 0 | 1
  Early Termination |  | 3.00 [3.0 to 3.0]

11. Secondary Outcome: ABC-2-C Domain Scores - Social Withdrawal
Description: The ABC-2 is an updated, empirically derived, validated 58-item caregiver-completed rating scale that measures the severity of a range of maladaptive behaviors commonly observed in children, adolescents, and adults with intellectual and developmental disabilities. The Community version of the scale (ABC-2-C) will be used. It is designed for use in individuals who are not residing in institutional settings. The checklist assesses symptoms across five domains: irritability, social withdrawal, stereotypic behavior, hyperactive/noncompliance, and inappropriate speech. Items are scored on a 4-point scale from 0 (never) to 3 (severe problem). The social withdrawal domain score range is 0-48, with higher scores indicating greater severity.
Time Frame: Baseline - Day 365, or early termination (prior to Day 365)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Baseline | 14.50 [11.0 to 18.0] | 16.00 [2.0 to 25.0]
  Day 28: number analyzed (Participants) | 2 | 3
  Day 28 | 7.50 [6.0 to 9.0] | 14.00 [7.0 to 17.0]
  Day 92: number analyzed (Participants) | 1 | 3
  Day 92 | 10.00 [10.0 to 10.0] | 12.00 [6.0 to 24.0]
  Day 183: number analyzed (Participants) | 1 | 1
  Day 183 | 10.00 [10.0 to 10.0] | 7.00 [7.0 to 7.0]
  Day 274: number analyzed (Participants) | 1 | 0
  Day 274 | 2.00 [2.0 to 2.0] |
  Day 365: number analyzed (Participants) | 1 | 0
  Day 365 | 4.00 [4.0 to 4.0] |
  Early Termination: number analyzed (Participants) | 0 | 1
  Early Termination |  | 22.00 [22.0 to 22.0]

12. Secondary Outcome: ABC-2-C Domain Scores - Stereotypic Behavior
Description: The ABC-2 is an updated, empirically derived, validated 58-item caregiver-completed rating scale that measures the severity of a range of maladaptive behaviors commonly observed in children, adolescents, and adults with intellectual and developmental disabilities. The Community version of the scale (ABC-2-C) will be used. It is designed for use in individuals who are not residing in institutional settings. The checklist assesses symptoms across five domains: irritability, social withdrawal, stereotypic behavior, hyperactive/noncompliance, and inappropriate speech. Items are scored on a 4-point scale from 0 (never) to 3 (severe problem). The stereotypic behavior subdomain score range is 0-21, with higher scores indicating greater severity.
Time Frame: Baseline - Day 365, or early termination (prior to Day 365)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Baseline | 8.00 [8.0 to 8.0] | 6.00 [0.0 to 15.0]
  Day 28: number analyzed (Participants) | 2 | 3
  Day 28 | 5.50 [5.0 to 6.0] | 13.00 [7.0 to 16.0]
  Day 92: number analyzed (Participants) | 1 | 3
  Day 92 | 6.00 [6.0 to 6.0] | 14.00 [8.0 to 15.0]
  Day 183: number analyzed (Participants) | 1 | 1
  Day 183 | 4.00 [4.0 to 4.0] | 6.00 [6.0 to 6.0]
  Day 274: number analyzed (Participants) | 1 | 0
  Day 274 | 8.00 [8.0 to 8.0] |
  Day 365: number analyzed (Participants) | 1 | 0
  Day 365 | 2.00 [2.0 to 2.0] |
  Early Termination: number analyzed (Participants) | 0 | 1
  Early Termination |  | 11.00 [11.0 to 11.0]

13. Secondary Outcome: ABC-2-C Domain Scores - Hyperactivity/Non-Compliance
Description: The ABC-2 is an updated, empirically derived, validated 58-item caregiver-completed rating scale that measures the severity of a range of maladaptive behaviors commonly observed in children, adolescents, and adults with intellectual and developmental disabilities. The Community version of the scale (ABC-2-C) will be used. It is designed for use in individuals who are not residing in institutional settings. The checklist assesses symptoms across five domains: irritability, social withdrawal, stereotypic behavior, hyperactive/noncompliance, and inappropriate speech. Items are scored on a 4-point scale from 0 (never) to 3 (severe problem). The hyperactivity/non-compliance subdomain score range is 0-45, with higher scores indicating greater severity.
Time Frame: Baseline until Day 365, or early termination (prior to Day 365)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Baseline | 32.00 [23.0 to 41.0] | 19.00 [13.0 to 38.0]
  Day 28: number analyzed (Participants) | 2 | 3
  Day 28 | 12.00 [6.0 to 18.0] | 22.00 [15.0 to 33.0]
  Day 92: number analyzed (Participants) | 1 | 3
  Day 92 | 40.00 [40.0 to 40.0] | 18.00 [14.0 to 35.0]
  Day 183: number analyzed (Participants) | 1 | 1
  Day 183 | 39.00 [39.0 to 39.0] | 18.00 [18.0 to 18.0]
  Day 274: number analyzed (Participants) | 1 | 0
  Day 274 | 40.00 [40.0 to 40.0] |
  Day 365: number analyzed (Participants) | 1 | 0
  Day 365 | 33.00 [33.0 to 33.0] |
  Early Termination: number analyzed (Participants) | 0 | 1
  Early Termination |  | 14.00 [14.0 to 14.0]

14. Secondary Outcome: ABC-2-C Domain Scores - Inappropriate Speech
Description: The ABC-2 is an updated, empirically derived, validated 58-item caregiver-completed rating scale that measures the severity of a range of maladaptive behaviors commonly observed in children, adolescents, and adults with intellectual and developmental disabilities. The Community version of the scale (ABC-2-C) will be used. It is designed for use in individuals who are not residing in institutional settings. The checklist assesses symptoms across five domains: irritability, social withdrawal, stereotypic behavior, hyperactive/noncompliance, and inappropriate speech. Items are scored on a 4-point scale from 0 (never) to 3 (severe problem). The inappropriate speech subdomain score range is 0-12, with higher scores indicating greater severity.
Time Frame: Baseline until Day 365, or early termination (prior to Day 365)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Units on a scale
  Baseline | 5.00 [2.0 to 8.0] | 2.00 [0.0 to 10.0]
  Day 28: number analyzed (Participants) | 2 | 3
  Day 28 | 1.50 [0.0 to 3.0] | 0.00 [0.0 to 2.0]
  Day 92: number analyzed (Participants) | 1 | 3
  Day 92 | 3.00 [3.0 to 3.0] | 0.00 [0.0 to 8.0]
  Day 183: number analyzed (Participants) | 1 | 1
  Day 183 | 1.00 [1.0 to 1.0] | 0.00 [0.0 to 0.0]
  Day 274: number analyzed (Participants) | 1 | 0
  Day 274 | 3.00 [3.0 to 3.0] |
  Day 365: number analyzed (Participants) | 1 | 0
  Day 365 | 2.00 [2.0 to 2.0] |
  Early Termination: number analyzed (Participants) | 0 | 1
  Early Termination |  | 0.00 [0.0 to 0.0]

15. Secondary Outcome: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to 52 weeks
Population: The safety analysis population is the same as the ITT population, assuming treatment is received as assigned at randomization.
Measure: Number; unit: Count of Participants
Arm/Group | Placebo | Basmisanil
Number analyzed (Participants) | 2 | 5
Count of Participants
  AEs | 2 | 5
  SAEs | 0 | 1

16. Secondary Outcome: Plasma Concentration of Basmisanil
Time Frame: Day 1 - Day 183
Population: The pharmacokinetic (PK) population consisted of all participants who received at least one dose of study treatment and who had data from at least one postdose sample. Only assessment time points with > 1 participant are shown due to concerns that certain demographic characteristics that may be present in only one treatment arm, or the duration a participant was in the trial, present an unacceptable risk of participant re-identification.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Basmisanil
Number analyzed (Participants) | 5
ng/mL
  Day 1 - Hour 1.5 | 2520 (965)
  Day 1 - Hour 3.5 | 2220 (955)
  Day 1 - Hour 5.5: number analyzed (Participants) | 4
  Day 1 - Hour 5.5 | 1640 (756)
  Day 1 - Hour 7.5: number analyzed (Participants) | 4
  Day 1 - Hour 7.5 | 1040 (392)
  Day 1 - Hour 9: number analyzed (Participants) | 3
  Day 1 - Hour 9 | 791 (368)
  Day 2 - Hour 0 | 731 (535)
  Day 2 - Hour 1.5: number analyzed (Participants) | 4
  Day 2 - Hour 1.5 | 2380 (576)
  Day 2 - Hour 3.5 | 2210 (864)
  Day 14 - Hour -1.5: number analyzed (Participants) | 2
  Day 14 - Hour -1.5 | 1210 (1230)
  Day 14 - Hour 0: number analyzed (Participants) | 4
  Day 14 - Hour 0 | 902 (973)
  Day 14 - Hour 1.5: number analyzed (Participants) | 4
  Day 14 - Hour 1.5 | 2480 (355)
  Day 14 - Hour 3.5 | 2160 (698)
  Day 92 - Hour 0: number analyzed (Participants) | 3
  Day 92 - Hour 0 | 896 (689)

17. Secondary Outcome: Plasma Concentration of the Basmisanil Metabolite M1
Time Frame: Day 1 - Day 183
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Basmisanil
Number analyzed (Participants) | 5
ng/mL
  Day 1 - Hour 1.5 | 1410 (585)
  Day 1 - Hour 3.5 | 1510 (417)
  Day 1 - Hour 5.5: number analyzed (Participants) | 4
  Day 1 - Hour 5.5 | 985 (335)
  Day 1 - Hour 7.5: number analyzed (Participants) | 4
  Day 1 - Hour 7.5 | 675 (221)
  Day 1 - Hour 9: number analyzed (Participants) | 3
  Day 1 - Hour 9 | 535 (173)
  Day 2 - Hour 0 | 664 (568)
  Day 2 - Hour 1.5: number analyzed (Participants) | 4
  Day 2 - Hour 1.5 | 1330 (358)
  Day 2 - Hour 3.5 | 1410 (506)
  Day 14 - Hour -1.5: number analyzed (Participants) | 2
  Day 14 - Hour -1.5 | 1400 (1410)
  Day 14 - Hour 0: number analyzed (Participants) | 4
  Day 14 - Hour 0 | 1060 (1470)
  Day 14 - 1.5: number analyzed (Participants) | 4
  Day 14 - 1.5 | 1510 (413)
  Day 14 - Hour 3.5 | 1250 (540)
  Day 92 - Hour 0: number analyzed (Participants) | 3
  Day 92 - Hour 0 | 648 (522)

18. Secondary Outcome: Quantitative EEG (qEEG) Beta-band Power
Description: This is the average of the EEG parameter 10 x Log_10 of the total beta power between 16 and 32 Hz in microVolt^2.
Time Frame: Baseline, Day 14
Measure: Mean (Standard Deviation); unit: µV2
Arm/Group | Basmisanil | Placebo
Number analyzed (Participants) | 2 | 5
µV2
  Baseline | 9.47 (0.21) | 11.39 (1.55)
  Day 14 | 9.44 (0.37) | 9.74 (1.05)

ADVERSE EVENTS:
Time Frame: Baseline - Day 365
Description: Observations where n </= 1 were combined into "unspecified" categories due to an unacceptable risk of participant re-identification.
Arm/Group | Placebo | Basmisanil
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/5
Other Adverse Events (participants affected / at risk) | 2/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | Basmisanil (N=5)
Unspecified SAE (General disorders) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | Basmisanil (N=5)
Incorrect dose administered (Injury, poisoning and procedural complications) | 2 (6) | 3 (7)
Unspecified AE (General disorders) | 1 (2) | 2 (7)

LIMITATIONS AND CAVEATS:
Data beyond certain timepoints (specified per outcome measure in the outcome measures section), or for timepoints for which n ≤ 1, is not reported due to concerns that certain demographic characteristics that may be present in only one treatment arm, or the duration a participant was in the trial, present an unacceptable risk of participant re-identification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT05307679/Prot_SAP_000.pdf